CLINICAL TRIAL: NCT06098391
Title: Results at More Than 10 Years of Meniscal Sutures Without Avivement
Acronym: SMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9060
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Knee Arthroscopy
Keywords: knee arthroscopy; Meniscal suture; Meniscal lesion; Meniscectomy; Arthroscopic suturing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, suturing the lesion is recommended rather than the classic meniscectomy, which leads to early and subsequent gonarthrosis. The most commonly practiced technique is arthroscopic suturing after avivement the area to be sutured to promote healing. But the real benefit of this enhancement has never been documented. The complexity of the surgical procedure makes the acceptability of this indication low by orthopedic surgeons at present (10% sutures compared to 90% meniscectomies).

The aim of the study is to evaluate the 10-year survival rate of meniscal sutures without avivement.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* Gender indifferent
* Patient operated on at the HUS between January 1, 2011 and June 30, 2013
* Medial or lateral meniscal lesion of the knee treated by arthroscopic suture without sharpening with or without reconstruction of the anterior cruciate ligament.
* Absence of written opposition in the medical file of the subject (and/or their legal representative if applicable) to the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Subject having expressed his opposition to the reuse of his data for scientific research purposes.
* Subject under judicial protection
* Subject under guardianship or curatorship
* Meniscal lesion not sutured or sutured with sharpening.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) having medial or lateral meniscal lesion of the knee treated by arthroscopic suture without avivement with or without reconstruction of the anterior cruciate ligament and operated on at the HUS between January 1, 2011 and June 30, 2013
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06-08 (Estimated)

PRIMARY OUTCOMES:
10-year survival rate of meniscal sutures without avivement | 10 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Orthopédie - Traumatologie Membre Supérieur - CHU de Strasbourg - France, Strasbourg, France